CLINICAL TRIAL: NCT05337293
Title: Coping in Heart Failure Partnership (COPE-HF): A Telephone-Based Intervention Study
Brief Title: Coping in Heart Failure Partnership Intervention
Acronym: COPE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: American Nurse Pracititioner Foundation (ANPF) (Unknown)
Responsible Party: Principal Investigator, Lucinda Graven, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015.14571
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: heart failure; problem-solving; social support; self-care
MeSH Terms: conditions — Heart Failure | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: This parallel 3-arm (intervention, attention, control) randomized controlled trial (N = 90) will concurrently enroll patients with heart failure to either a 12-week intervention (COPE-HF Partnership), a 12-week attention group (contacts spaced similarly to that of the intervention group), or a control group. All data collection contacts occur at identical intervals among groups.
Who Masked: Outcomes Assessor
Masking Description: All data were collected by a research assistant blinded to study group assignment and purpose of study. A second research assist blinded to study purpose and intervention conducted all participant contacts with the attention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPE-HF Partnership Intervention (Experimental): Working with a trained registered nurse interventionist, participants in this arm were trained to use a 4-step problem-solving process to manage identified problems related to heart failure. Heart failure self-care education and materials were provided as indicated based on specific identified problems.
  Interventions: Behavioral: COPE-HF Partnership Intervention
- Attention (Sham Comparator): Participants in this arm received telephone calls from a trained research assistant on the same schedule as the intervention group. During these calls basic data were collected on several key areas of heart failure self-care. No intervention or patient education took place during these calls.
  Interventions: Other: Attention
- Usual Care (No Intervention): Participants in this arm received usual care from their healthcare providers and facility designated heart failure discharge education only.

INTERVENTIONS:
Behavioral: COPE-HF Partnership Intervention — Participants were trained to use a 4-step problem-solving process based on the Theory of Social Problem-Solving (TSPS) to manage HF-related problems experienced in the home over 12-weeks. The core belief of TSPS is effective problem-solving requires a positive problem orientation (i.e., viewing problems as a challenge versus a threat) and elicits rational problem-solving versus avoidance or impulsivity/carelessness. Problem-solving follows from a positive problem orientation and involves accurate problem identification, generation of appropriate potential solutions, active decision-making, and solution implementation and evaluation. The goal of this intervention was to move HF patients toward a positive problem orientation and use of rational problem-solving strategies that support greater HF self-care and reduce depression. The COPE-HF Partnership Intervention consisted of 1 home visit and 7 follow-up telehealth sessions led by a registered nurse interventionist.
  Arms: COPE-HF Partnership Intervention
Other: Attention — Participants in the attention group received a sham intervention that consisted of scheduled telephone calls consistent with the timing of that received by the intervention group. During these calls, basic information was gathered on key areas of heart failure self-care management and the frequency of healthcare usage. No intervention or education was provided.
  Arms: Attention

SUMMARY:
The purpose of this study is to examine the feasibility and preliminary effectiveness of a 12-week support and problem-solving telephone-based intervention (COPE-HF) on heart failure self-care, depression, and healthcare utilization. Heart failure patients will be randomized to one of three groups (intervention, attention, control), with data collected at baseline and at 5, 9, and 13 weeks.

DETAILED DESCRIPTION:
The long-term goal of this research is to reduce morbidity and improve heart failure self-care and depression in heart failure patients. The initial step in meeting this goal is to pilot-test a telephone-based, tailored support and problem-solving intervention (COPE-HF Partnership) to improve HF self-care and depression in a sample of heart failure patients. The following research aims are to: 1) test the COPE-HF Partnership intervention and determine its feasibility and acceptability for managing HF-related problems; and 2) evaluate the preliminary effects of the COPE-HF Partnership intervention on heart failure self-care, depression, and healthcare utilization. This study will be guided by quantitative methods and include a repeated measures, randomized controlled trial to evaluate the feasibility, acceptability, and preliminary effectiveness of the 12-week COPE-Partnership intervention in a sample of heart failure patients (n = 90). Participants for this study will be recruited from from the cardiac/telemetry floors at Tallahassee Memorial Hospital and Capital Regional Medical Center in Tallahassee, FL.

The target recruitment size was 90 participants based upon attrition rates reported in previous studies (35%) and the number of participants needed to provide trend data in preparation for a larger, more adequately powered clinical trial. Following verbal informed consent, all participants were screened for cognitive impairment using the 6 Item Cognitive Impairment Test (6CIT) prior to baseline data collection. Data were collected using the following instruments: a Sociodemographic and Clinical Survey (baseline only), the Self-Care of HF Index (SCHFI; v. 6.2), the Heart Failure Symptom Survey (HFSS), the Interpersonal Support Evaluation List-12 (ISEL-12), the Social Problem-Solving Inventory Revised (SPSIR), Healthcare Utilization Survey, the Center for Epidemiological Studies-Depression (CESD), the Family APGAR.

Participants randomized to the intervention group participated in a telephone-based support and problem-solving training intervention over 12 weeks (Weeks 1-4, 6, 8, 10, 12).

Participants randomized to the attention group received usual care plus telephone calls on the same schedule as the intervention group and consisted of a health check with information collected regarding recent healthcare usage.

Participants randomized to the control group received usual care from their healthcare providers and received heart failure self-care education upon discharge from the healthcare facility.

Follow-up data collection occurred at weeks 5, 9, 11, 13. All data were self-report and collected by a trained research assistant who collected study data over the telephone and marked participants answers on a computerized data spreadsheet. Data were analyzed using linear and multi-level modeling approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a primary or secondary diagnosis of HF
2. Undergoing medical treatment for HF
3. BNP >100
4. Able to read, speak, and understand English
5. Reliable telephone access
6. Live within 100 miles of acute care facility

Exclusion Criteria:

1. Diagnosis of heart failure due to a correctable cause or condition
2. Reduced life expectancy < 12 months
3. History of cognitive impairment or a score >8 on the 6CIT
4. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Self-care Maintenance | baseline, 5 weeks
  Self-care maintenance was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Maintenance | baseline, 9 weeks
  Self-care maintenance was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Maintenance | baseline, 13 weeks
  Self-care maintenance was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Management | baseline, 5 weeks
  Self-care management was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Management | baseline, 9 weeks
  Self-care management was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Management | baseline, 13 weeks
  Self-care management was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Confidence | baseline, 5 weeks
  Self-care confidence was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Confidence | baseline, 9 weeks
  Self-care confidence was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-care Confidence | baseline, 13 weeks
  Self-care confidence was self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.

SECONDARY OUTCOMES:
Depression | baseline, 5 weeks
  Depression was self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Depression | baseline, 9 weeks
  Depression was self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Depression | baseline, 13 weeks
  Depression was self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Healthcare utilization | baseline, 5 weeks
  Healthcare utilization was determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.
Healthcare utilization | baseline, 9 weeks
  Healthcare utilization was determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.
Healthcare utilization | baseline, 13 weeks
  Healthcare utilization was determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.

OTHER OUTCOMES:
Heart Failure Symptoms | baseline, 5 weeks
  Symptoms of HF were assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | baseline, 9 weeks
  Symptoms of HF were assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | baseline, 13 weeks
  Symptoms of HF were assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Social Problem-Solving | baseline, 5 weeks
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Social Problem-Solving | baseline, 9 weeks
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Social Problem-Solving | baseline, 13 weeks
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Social Support | baseline, 5 weeks
  Social support was self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.
Social Support | baseline, 9 weeks
  Social support was self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.
Social Support | baseline, 13 weeks
  Social support was self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda J Graven, PhD APRN, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Capital Regional Medical Center, Tallahassee, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.